CLINICAL TRIAL: NCT05511168
Title: Craniosynostosis : Surgical Treatment Modalities and Outcome
Brief Title: Craniosynostosis :Surgical Treatment Modalities and Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Amgad Kotb, Craniosynostosis: surgical treatment modalities and outcome, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Craniosynostosis:outcome
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Craniosynostoses
Keywords: Surgical treatment modalities and outcome
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Craniosynostosis patients (Other): Craniosynostotic patients aged more than 3months
  Interventions: Procedure: Craniostnostosis surgery

INTERVENTIONS:
Procedure: Craniostnostosis surgery — Surgery of craniosynostosis

SUMMARY:
Aim of study:

1. To evaluate outcome of cases( cosmoses and cognition) after Craniosynostosis surgery
2. - To ascertain intra- and postoperative complications

DETAILED DESCRIPTION:
Craniosynostosis is defined as the premature fusion of one or more of the sutures normally separating the infant's skull bony plates, resulting in abnormal growth of the cranial vault and skull base, which may influence brain growth and development(1).

Aetiology Primary Craniosynostosis: No cause for the synostosis is recognized in the majority of cases, , but in an increasing proportion (currently about 25%), a mutation is identified. A considerable proportion of these mutations are related to six genes FGFR2, FGFR3, TWIST1, EFNB1, TCF12 and ERF(2).

Types of Craniosynostosis Non-syndromic (or isolated), in which only the skull is affected, The syndromic craniosynostosis is caused by an inherited or genetic condition and associated with craniofacial syndromes(3).

Syndromic craniosynostosis is most commonly found in:

* Apert syndrome
* Crouzon syndrome
* Muenke syndrome
* Pfeiffer syndrome
* Saethre-Chotzen syndrome(4)

Diagnosis:

The skull shape from all directions, and the measurement of the head circumference for calculating the cephalic index (the ratio of maximum breadth to maximum length of the skull). Any sutural ridging, prominent blood vessels on the scalp, and the size, shape and tension of the fontanels should also be assessed.

For evaluating ICP, ophthalmological examination is of great importance. In cases with increased ICP, papilledema is present To confirm the diagnosis The computed tomography (CT) with three-dimensional (3D) reconstruction is considered the most complete and accurate imaging to diagnose craniosynostosis the magnetic resonance imaging (MRI) is an excellent technique for the evaluation of brain(5).

Many types of craniosynostosis require surgery. The surgical procedure is done to relieve pressure on the brain, correct the craniosynostosis, and permit the brain to grow appropriately. Babies with very mild craniosynostosis might not need surgery. Delay surgical intervention causes irreversible loss of vision and permanent cognitive impairment.

a neglected case of craniostenosis, presented with deformity of head with mental retardation, which was operated after delay lead to poor neurological outcome(6).

Surgical management for craniosynostosis is based on the suture(s) involved, the age of the child, and the individual needs for each patient.

* Strip craniectomy
* Sagittal springs also known as cranial spring surgery
* Fronto-orbital advancement /reshaping
* Cranial vault remodeling and reconstruction.
* Posterior vault distraction osteogenesis (7) Outcome variables debated include magnitude and durability of head shape improvement, cost, neurodevelopmental trajectory, burden of care to patient, and intra- and postoperative complication rates(8).

Most frequent complication was non-filiated postoperative hyperthermia followed by infection , subcutaneous haematoma), dural tears and cerebrospinal fluid (CSF) leakage. Number and type of complications was higher among the group of reoperated patients (9).

ELIGIBILITY:
Inclusion Criteria:

* all patients either syndromic or nonsyndromic

Exclusion Criteria:

* • Patients aged less than 3 month

  * Patients had bad general condition

Ages: 3 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Cosmosis | 1 year
  cosmosis of patients after Craniosynostosis surgery by these measures : Cephalic index

SECONDARY OUTCOMES:
intraoperative bleeding | 1 year
  Volume of blood lost in the operation